CLINICAL TRIAL: NCT00371553
Title: Prospective Open-Labeled Non Randomised Phase-II Study of SU011248 (Sunitinib) in Male Patients With Relapsed or Cisplatin-Refractory Germ Cell Cancer - A CUOG / GTCSG Cooperative Phase II Study -
Brief Title: Phase-II Study of SU011248 (Sunitinib)in Male Patients With Relapsed or Cisplatin-Refractory Germ Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Canadian Urologic Oncology Group (Other); NCIC Testis Group (Unknown); German Testicular Cancer Study Group (Other)
Responsible Party: Dr Christian Kollmannsberger, BC Cancer Agency
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Testis protocol Version 003; CUOG-TE 05/OZM-007
Record Dates: First submitted 2006-09-01; First posted 2006-09-04 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2009-07

CONDITIONS: Relapsed or Cisplatin-Refractory Germ Cell Cancer
Keywords: relapsed or cisplatin-refractory germ cell cancer; germ cell cancer; SU011248 (Sunitinib)
MeSH Terms: conditions — Recurrence; Neoplasms, Germ Cell and Embryonal | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: SU011248 (Sunitinib)

SUMMARY:
The purpose of this study is to investigate the activity of SU011248 in subjects with cisplatin-refractory or multiply relapsed germ cell cancer. It is believed that SU011248 treatment may prove to increase disease response.

DETAILED DESCRIPTION:
SU011248 is a new investigational drug that has been shown to be effective against kidney cancer and other cancers in clinical trials. An investigational drug in Canada is a drug that is not yet approved for standard treatment. SU011248 inhibits enzymes (chemicals that help cells function) called tyrosine kinases, which are important enzymes for tumor growth and tumor spread in your body. If these enzymes are blocked, tumor growth may be disrupted and subsequently the cancer cell may die. SU011248 has been given to patients with kidney cancer and other cancers in clinical trials and some of them have improved, although it is not yet certain how often this occurs. There is some evidence that the enzymes inhibited by SU011248 also play an important role in the development and growth of germ cell cancers. This is the reason why SU011248 is being tested in subjects with germ cell cancers.

Objectives:

Primary:

To assess the response rate of SU011248 in patients with relapsed or cisplatin- refractory germ cell cancer.

Secondary: To assess the rate of disease stabilizations, toxicity, time to progression and response duration of SU011248 given to patients with relapsed or cisplatin-refractory germ cell cancer.

Study Drug Regimen:

SU011248 will be given at 50 mg once daily for 4 consecutive weeks followed by a 2-week rest period to comprise a complete cycle of 6 weeks. SU011248 will be orally self-administered once daily without regard to meals. Patients will remain on the study drug until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* patients with histologically proven seminomatous or non-seminomatous germ cell cancer
* patients with relapse within 8 weeks after at least 2 different cisplatin- based regimens or
* patients with disease progression or relapse after salvage high-dose chemotherapy or patients with disease progression during cisplatin-based chemotherapy or patients with contraindications for other aggressive chemotherapy
* measurable disease
* Life expectancy of greater than 3 months
* Karnofsky Performance status > 60
* age > 18
* adequate organ function
* Resolution of acute toxic effects of prior radiotherapy, surgical procedure or chemotherapy to NCI CTCAE Version 3.0 <= grade 1.
* Left ventricular ejection fraction (LVEF) >= lower limit of normal (LLN) as defined by the institution performing the scan as assessed by multigated acquisition (MUGA) scan or echocardiography
* Signed and dated informed consent document
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* Acute infection
* Uncontrolled intercurrent illness
* Patients with a history of other active malignancy in the past 5 years (with the exception of adequately treated cervical carcinoma in situ and non melanomatous skin cancers) are excluded.
* Interval from last chemotherapy < 3 weeks.
* Simultaneous radiation of the only target lesion
* NCI CTCAE grade 3 hemorrhage < 4 weeks of starting the study treatment
* Patients must not be on therapeutic anticoagulation.
* Major surgery or radiation therapy within < 4 weeks of starting the study treatment.
* History of or known brain metastases, spinal cord compression, or carcinomatous meningitis, or evidence of brain or leptomeningeal disease
* Any of the following within the 12 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism.
* Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication.
* Ongoing cardiac arrhythmias of NCI CTCAE grade >= 2, atrial fibrillation of any grade, or prolongation of the QTc interval to >500 msec on baseline EKG.
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
* Hypertension that cannot be controlled by medications (>150/100 mm Hg despite optimal medical therapy).
* Current treatment on another clinical trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2006-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Response Rate

SECONDARY OUTCOMES:
Rate and duration of stable disease
Time to progression.
Median and 1 yr survival
Safety and tolerability of SU011248

CONTACTS AND LOCATIONS:
Overall Officials: Christian K Kollmannsberger, MD, Principal Investigator — BC Cancer Agency -Vancouver Centre
Locations (6):
- Canada (6):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - BC Cancer Agency - Vancouver Centre, Vancouver, British Columbia
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - QEII Health Science Center, Halifax, Nova Scotia
  - London Regional Cancer Centre, London, Ontario
  - Princess Margaret Hospital, Toronto, Ontario